CLINICAL TRIAL: NCT04367623
Title: Exploring Brain Computer Interface Controlled Functional Electrical Stimulation as a Motor Conditioning Strategy Prior to Physical Practice in People With Subacute Spinal Cord Injury
Brief Title: Motor Conditioning to Enhance the Effect of Physical Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays in approval process, COVID restrictions, staffing shortages
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN19NE396
Record Dates: First submitted 2020-02-13; First posted 2020-04-29 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients receiving conventional hand therapy, time matched to the duration of total intervention in the Active group
  Interventions: Other: Brain computer interface based therapy
- Active (Active Comparator): Patients receiving BCI FES prior to the conventional therapy
  Interventions: Other: Brain computer interface based therapy

INTERVENTIONS:
Other: Brain computer interface based therapy — Participants who decide to take part will be assigned to a treatment or a control group. Both groups will have the same assessments and the same number of therapy sessions. Therapy group will have a training that consists of Brain Computer Interface controlled Functional Electrical Stimulation followed by a physical practice of the dominant upper limb, while the control group will have a physical practice only. One experimental session will last about 60 min for both groups (including setup and therapy) and participants in each group will receive 20 sessions, about 3 times per week. The expected time needed for completion of 20 sessions is 7 weeks

SUMMARY:
Spinal Cord Injury (SCI) affects person's ability to move and feel sensation from the body. About half of patients with tetraplegia (high level SCI) have an incomplete injury, i.e. have some sensation and control of muscles preserved and could recover some function of their upper limbs. In this study the researchers would like to increase the effect of physical therapy of the upper limbs by sensory-motor priming. To achieve this they will use Brain Computer Interface (BCI) controlled Functional Electrical Stimulation (FES) immediately prior to the physical therapy of the upper limbs. BCI will be operated by motor attempt (motor priming) which will activate the FES applied to participants' hand muscles to achieve movement (sensory and motor priming). Physical therapy in this study will not replace conventional therapy that participant receive as a part of their standard treatment. There will be two groups: a treatment group (BCI FES with physical therapy) and a control group (physical therapy only), each receiving 20 therapy sessions of matched duration (40-50 min) of their dominant hand. Based on power analysis and results from our study (Osuagwu et al. 2016, J Neural Eng) there will be thirteen participants per group matched by age and the level of injury. Therapy will be applied to dominant hand only, because of the limited time available for experimental studies on participants who are already under active rehabilitation programme. Primary measures will be functional outcomes (range of movement, muscle strength, grip force, independence) while secondary outcomes will be neurological outcomes (EEG activity) and quality of life measures. The outcomes will be compared between the treatment and the control group and between the dominant and the non-dominant hand of each participant.

DETAILED DESCRIPTION:
Participants who decide to take part will be assigned to a treatment or a control groups. Both groups will have the same assessments and the same number of therapy sessions. Therapy group will have a training that consist of Brain Computer Interface controlled Functional Electrical Stimulation followed by physical practice of the dominant upper limb while the control group will have physical practice only. One experimental session including will last about 60 min for both groups (including setup and therapy) and participants in each group will receive 20 sessions, about 3 times per week.

1. Assesments There will be three assessments: an initial assessment within a week prior to the first therapy session, a final assessment within a week following the last therapy session and a follow up session 3 months after the last therapy session. Assessments will consist of qualitative and quantitative measures. It will comprise of assessments of motor functions, neurological functions and participants feedback on the therapy (questionnaires and. Interviews)
2. Therapy There will be 20 therapy sessions for each group 2.1. Therapy Treatment Group This will consist of 30 min of BCI FES followed by 30 min of physical practice of the dominant upper limb. We decided to include only dominant arm/hand from two reasons: Each participant can be their own control to compare the outcome between hands. The other reason is that it is not possible to find more than an hour free time in between of their regular physical therapies and other activities. 2.1.1. BCI FES Participants will be wearing an EEG device (Epoch, Emotiv) and will have several pair of self-adhesive FES electrodes attached to their arms, over muscles that control reaching and grasping. The exact location and number of FES electrodes will be patient specific and will depend on their functional ability.

Each therapy session will start with a 5 min long calibration (to set BCI parameters for that day) followed by training.

During calibration phase participants will watch a computer screen showing a hand squeezing a ball. Participants will imagine doing the same action while their EEG will be recorded. BCI-FES Upon seeing a visual cue (a small cross) on a screen, participants attempt to move their dominant arm and hand to achieve reach and grasp movement towards an object (e.g. a plastic bottle). They repeat this 30 to 40 times in total, targeting 30 successful trials. The number of trials is based on our previous study (Osuagwu et al 2016, J Neural Eng). During each trial, upon the appearance of cue on the screen, the participant has 10 seconds to attempt movement to activate FES. They will practice movements of one hand only so there will be only one type of cue. On a successful attempt, FES will be initiated for 10-15 seconds to complete reach and grasp movement. An anti-gravity support will be used to assist movement, if necessary. This might be mentally demanding for some participants, and they might require breaks in between trials. Thus although BCI FES effectively lasts about 10 min (the same as in our previous study) the whole BCI FES session will take about 30 min. BCI FES will be immediately followed by physical practice. It is not possible to wait for participants regular occupation therapy because of a relatively short duration of the motor priming effect (from the literature it is 10-30 min).

After 1st, 5th, 10th , 15th and 20th session participants will fill out NASA task load index questionnaire, which takes about 5 min. This measures their workload. 2.1.2. Physical practice Immediately after BCI FES, participant will have physical therapy for 30 min. The objects and devices typically used in occupational therapy, putty, pegboards, nut-bolt-boards, rings, etc will be used for reaching and grasping tasks. These tasks may change over time depending on the capability of participant. FES will not be used in this phase 2.2. Therapy Control Group Control group will receive 40 min of physical practice only, that will be similar to the physical practice in the treatment group. Total duration is based on the total duration of BCI FES (10 min) and physical practice (30 min) in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Upper and lower age limit as above
2. Incomplete spinal cord injury at level C3-C8 or complete spinal cord injury (C3-C8) with a zone of partially preserved innervation
3. Sub-acute patients, likely to remain as inpatient during the period of study
4. Normal or corrected to normal vision

Exclusion Criteria:

1. Self reported neurological conditions prior to the injury that are expected to substantially change the EEG signal (e.g. stroke, epilepsy, brain injury, Parkinson's disease)
2. Inability to understand the experimental task
3. Brain, brachioplexus or peripheral nerve damage occurring at the time of the spinal cord injury.
4. General contraindications for using FES (implanted devices, pregnancy, sensitive skin, automatic dysreflexia)
5. Halos (large neck supports surrounding head) preventing EEG recording
6. Inability to sit for 1.5 hour due to skin redness or sores
7. Infections and general poor health due to injury
8. Unable to speak English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in Spinal Cord Independence measure (range 0 to 100, max 100) | two months: baseline and upon completion of the therapy, typically 9 weeks
  Spinal Cord Independence measure Questionnaire regarding independence in activities of daily living
Change in the hand range of motion (range 0 to 90 degress, max 90 degress) | two months: baseline and upon completion of thetherapy, typically 9 weeks
  Change in the range of motion measured by goniometer (o degrees)
Changes in the Manual muscle test (range 0 to 5, max 5) | two months: baseline and upon completion of the therapy, typically 9 weeks
  Change of strength of individual hand and arm muscles
Change in grip strength (range 0 to 80 N, max 80 N) | two months: baseline and upon completion of the therapy, typically 9 weeks
  Change in grip strength (N)

SECONDARY OUTCOMES:
Changes in Multichannel brain activity measured by electroencephalography (EEG) during attempted or imagined movements | two months: baseline and after completion of the therapy, typically 9 weeks
  Event related synchronisation/desynchronsation (%) (-200% to 100%, max 100%)
Changes in baseline multichannel electroencephalogaphy (EEG) measurement | two months: baseline and upon completion of the therapy, typically 9 weeks
  Measurement of brain activity at rest (%) (0-100%, max 100%)
Changes NASA (National Aeronautics and Space Administration) task load index | after 1st, 10st and 20th therapy session (typically 0, 3 and 9 weeks -there is a washout peiord between first and last 10 sesions)
  Questionnaire measuring mental work load during therapy (0 very low to 10 very high)
Quebec User Evaluation of Satisfaction with Assistive Technology | Upon completion of the therapy, typically 9 weeks
  questionnaire (two parts. Part 1 Device range 0 to 40, max 40; Part 2 Services, range 0 to 20, max 20)
Patient feedback, satisfaction with therapy | Upon completion of the therapy, typically 9 weeks
  semistructured interview (no units)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Vuckovic, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osuagwu BC, Wallace L, Fraser M, Vuckovic A. Rehabilitation of hand in subacute tetraplegic patients based on brain computer interface and functional electrical stimulation: a randomised pilot study. J Neural Eng. 2016 Dec;13(6):065002. doi: 10.1088/1741-2560/13/6/065002. Epub 2016 Oct 14. PMID 27739405